CLINICAL TRIAL: NCT00212667
Title: Controlled Study of ONO-5920 in Patients With Involutional Osteoporosis in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-5920-02; NCT00189891 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Involutional Osteoporosis
Keywords: ONO-5920, osteoporosis, bisphosphonate
MeSH Terms: conditions — Osteoporosis | interventions — YM 529

INTERVENTIONS:
Drug: ONO-5920

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-5920 in patients with involutional osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with fragility fracture according to the diagnostic criterial for the diagnosis of Primary Osteoporosis
2. Patients having radiographically confirmed vertebral (T4-L4) fractures
3. Other inclusion criteria as specified in the study protocol

Exclusion Criteria:

1. Patients having secondary osteoporosis or another condition that presents low bone mass
2. Patients having findings on X-ray that affect evaluation of vertebral fracture
3. Patients that have been administered bisphosphonate derivatives
4. Other exclusion criteria as specified in the study protocol

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2002-08; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
New fragility vertebral fracture

SECONDARY OUTCOMES:
New clinical fracture, biochemical markers of bone turnover, height, mean bone mineral density of the lumbar spoine (L2-4 BMD), lower back pain

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. LtTd.

REFERENCES:
- [Derived] Matsumoto T, Hagino H, Shiraki M, Fukunaga M, Nakano T, Takaoka K, Morii H, Ohashi Y, Nakamura T. Effect of daily oral minodronate on vertebral fractures in Japanese postmenopausal women with established osteoporosis: a randomized placebo-controlled double-blind study. Osteoporos Int. 2009 Aug;20(8):1429-37. doi: 10.1007/s00198-008-0816-7. Epub 2008 Dec 20. PMID 19101754